CLINICAL TRIAL: NCT06301451
Title: Efficacy and Safety of Portable Hydrogen Rich Water Machine is Used for Adjuvant Treatment of Patients With Hyperlipidemia: #A Prospective, Multicenter, Follow-up Machine-controlled, Standard-controlled Clinical Trials
Brief Title: Efficacy and Safety of Portable Hydrogen Rich Water Machine is Used for Adjuvant Treatment of Patients With Hyperlipidemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Jia (Other)
Responsible Party: Sponsor-Investigator, Sun Jia, Vice-Chairman of the Department of Endocrinology and Metabolism#Chief Physician#Associate Professor#Doctor Supervisor of Endocrinology, Zhujiang Hospital
Organization: Zhujiang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XD2021-1
Record Dates: First submitted 2022-03-30; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Hyperlipidemias
Keywords: Hydrogen; Hydrogen rich water; Efficacy and safety; Adjuvant therapy
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: It is estimated that 180 subjects will be enrolled and randomly divided into the experimental group and the control group according to 2:1. During the observation period, the experimental group drink the hydrogen water prepared by the experimental equipment on the basis of the general dietary guidance, while the control group adopted the general dietary guidance. Every subject's diet and lifestyle remains largely unchanged during the treatment period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General dietary guidance and hydrogen water group (Experimental): Trial group is treated with general dietary guidance and hydrogen water prepared by portable hydrogen rich water machine.
  Interventions: Device: General dietary guidance and hydrogen water prepared by portable hydrogen rich water machine
- General dietary guidance group (No Intervention): Control group is treated with general dietary guidance.

INTERVENTIONS:
Device: General dietary guidance and hydrogen water prepared by portable hydrogen rich water machine — The trial group drink the hydrogen water prepared by the experimental equipment on the basis of receiving general dietary guidance.
  Arms: General dietary guidance and hydrogen water group

SUMMARY:
In the past 30 years, the blood lipid level of the Chinese population has gradually increased, and the prevalence of dyslipidemia patients has increased significantly. Hyperlipidemia is a disease caused by abnormal blood lipid levels, also known as abnormal lipid metabolism. Common clinical indicators include total cholesterol (TC), triglyceride (TG), low-density lipoprotein (LDL) and high-density lipoprotein ( HDL).The number of patients with abnormal blood lipid levels in China accounts for as high as 40% of the total. It is estimated that between 2010 and 2030,cardiovascular disease events will increase by 9.2 million, which seriously endangers human health and becomes a high risk factor for various cardiovascular diseases, such as atherosclerosis. One of the pathological foundations of atherosclerosis is that abnormal lipid levels in the body cause a large amount of lipid to be deposited in the arterial endothelial matrix, which is phagocytosed by smooth muscle and macrophages to form foam cells.

Hydrogen, the lightest and smallest molecular gas in the atmosphere, is considered a novel antioxidant that reduces oxidative stress. Accumulating evidence from various biomedical fields in clinical studies and experimental models of many diseases suggests that hydrogen inhalation or drinking hydrogen-containing solutions can be used as a therapeutic strategy. Due to the special physical properties of hydrogen gas that is easy to diffuse, hydrogen molecules can penetrate cell membranes to reach organelles and cell nuclei. Hydrogen's moderate reducing properties make it effective in reducing cytotoxicity, protecting nuclear DNA and mitochondria, and reducing the risk of lifestyle-related diseases and cancer.

In addition, hydrogen intake can reduce oxidative stress, improve cellular function, and reduce chronic inflammation, which are associated with the pathology and etiology of hyperlipidemia and other related diseases. Molecular hydrogen can regulate important metabolic functions such as signal transduction, protein phosphorylation, miRNA expression, and autophagy. Studies have shown that intake of hydrogen water in APOE knockout mice can reduce serum total cholesterol and low-density lipoprotein levels and prevent the progression of atherosclerosis. A study by Song et al. in 2013 included 20 subjects who drank 0.9 to 1 L of hydrogen-rich water per day for 10 weeks, and the subjects' LDL-C levels decreased significantly before and after treatment. Another study showed that subjects with underlying lipid metabolism abnormalities were treated with high-concentration hydrogen water (5.5mmol/d) for up to 24 weeks, and serum total cholesterol and low-density lipoprotein levels were significantly reduced. Protein function and redox status (eg, increased serum superoxide dismutase and decreased malondialdehyde) were improved, markers of inflammation (eg, serum tumor necrosis factor-alpha) decreased and fasting blood glucose decreased. At present, the research on the treatment of hyperlipidemia with hydrogen water is very limited. The portable hydrogen water hydrogen machine used in this study has passed the registration test of the Guangdong Provincial Medical Device Quality Supervision and Inspection Institute. In order to evaluate the use of the portable hydrogen water hydrogen machine for hyperlipidemia The efficacy and safety of adjuvant therapy in patients, this clinical trial is specially carried out.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized, standard-controlled clinical trial with an expected enrollment of 180 subjects. The subjects who meet the conditions of this trial will be randomly divided into the experimental group and the control group according to 2:1. The experimental group drank hydrogen water prepared by the experimental device on the basis of general dietary guidance, while the control group only received general dietary guidance, and the diet and lifestyle of each subject remained basically unchanged during the treatment period. This clinical trial is equipped with a nutritionist, who will provide general dietary guidance to the subjects before the formal trial. The subjects in the experimental group also need to receive additional training on the use of experimental equipment. During the research process, subjects need to fill in the online electronic diary card 3 days a week (2 days on weekdays and 1 day on weekends), and take photos and upload the diet on the day, and the dietitian will monitor the subjects' diet every week. Evaluate and give guidance; high-fat and high-sugar foods during the trial period need to be specially recorded in the electronic diary card, and daily hydrogen water intake, weekly tobacco, alcohol intake and physical activity are also recorded in the electronic diary card. On the 14th day of the treatment period, the subjects in the experimental group were followed up by telephone, mainly to investigate the use of the experimental equipment. At 1 month, 3 months, and 6 months after the start of treatment, the subjects returned to the hospital for follow-up, received corresponding laboratory tests, and evaluated the triglyceride levels of the experimental group and the control group at 1 month, 3 months, and 6 months. Absolute and percent change from baseline in lipids, total cholesterol, HDL cholesterol, LDL cholesterol, non-HDL cholesterol, small and dense LDL, apolipoprotein B, TNF-alpha , to study product performance, as well as adverse events during treatment, serious adverse events, and device defects to evaluate the efficacy and safety of portable hydrogen water hydrogen generators.

The statistical methods are as follow:

1.General Principles of Statistical Analysis:

1. Test standard: α=0.05 two-sided test is adopted uniformly, and P≤0.05 is considered to be statistically significant.
2. Measurement data: We use mean ± standard deviation to represent measurement data, and if necessary, give data such as minimum value, maximum value, P25, median and P75. When comparing before and after treatment between or within the two groups, the variables are first tested for normality. When obeying normal distribution, use group t-test or paired t-test; when obeying non-normal distribution, use nonparametric statistical methods such as Wilcoxon rank sum test or Signed Rank test. If the influence of center or other factors is considered, use analysis of covariance.
3. Count data: We use the frequency and its percentage to statistically describe the count data. The chi-square test, Fisher's exact test or Wilcoxon rank-sum test are used for comparison between two groups or within groups before and after treatment; if the influence of center or other factors is considered, the CMH chi-square test adjusted for center effect was used.
4. Subgroup analysis: We do not exclude subgroup analyses when necessary.

2.Statistical analysis crowd:

1. Full Analysis Set, FAS: The full analysis set is obtained by including all randomized subjects as much as possible according to the intention-to-treat principle. All patients who receive at least one therapeutic intervention and had at least 1 post-intervention efficacy evaluation data (at least 1 LDL-C, TG, TC, HDL-C data at month 1, 3 or 6) should be included in the full analysis set.
2. Per Protocol Set，PPS: Refers to all subjects who completed the trial and excluded serious protocol violations. The PPS population includes the FAS population who meet the following criteria: ①Compliance with drinking hydrogen water: During the trial period, subjects drink 8 cups of hydrogen water per day according to the protocol, a total of 1200mL; ②There is no major violation of the protocol, such as taking prohibited drugs specified in the protocol; ③No major evaluation indicators are missing, and so on.
3. Safety Analysis Set，SS: All subjects who receive at least one therapeutic intervention and have data on at least one post-intervention safety assessment.

3.Demographic and Baseline Statistical Comparison: We use the FAS set to statistically describe the subjects' demographic data (gender, age, height, weight) and baseline data, and test their balance between the experimental and control groups. Among them, the mean, standard deviation, minimum value, maximum value, median, 25th percentile and 75th percentile are described by measurement data; frequency and corresponding percentage are described by count data; count data are described by chi-square test or Fisher's exact test; nonparametric tests for quantitative indicators using independent t-test or Wilcoxon two-sample test.

4.Statistical comparison of efficacy indicators:

1. Primary efficacy indicator: In this study, the FAS set and the PPS set were used to compare the main evaluation index, the percentage change from baseline in low-density lipoprotein cholesterol (LDL-C) after 3 months of treatment, between the experimental group and the control group, respectively. A mixed-effects model with repeated measures (MMRM) was used, with treatment group, trial center, visit, and treatment group-visit interaction terms as fixed factors, baseline measurements as covariates, and unstructured covariances. The matrix models the within-subject correlations. The denominator degrees of freedom are calculated using the Kenward-Rogers approximation. If the above model fails to converge, assume heterogeneous Toeplitz and heterogeneous first-order autoregressive Toeplitz in turn. The first covariance structure that yields convergence is used for analysis. The primary analysis of the primary efficacy endpoint will be based on observational data only, with no imputation for missing data. We calculate the difference and 95% confidence interval of the least square means of the two groups. If the upper limit of the 95% confidence interval of the difference of the least square means of the main indicators is less than 0%, it means that the experimental group is superior to the control group.Covariance (ANCOVA) model is used to conduct the sensitivity analysis of the main evaluation indicators, and the percentage of changes in low-density lipoprotein cholesterol (LDL-C) relative to the baseline in the third month of the main evaluation index is compared between the experimental group and the control group, respectively. For comparison, missing data are imputed using LOCF. Baseline measurements are used as covariates, and treatment group and study center were fixed effects. Calculate the difference and 95% confidence interval of the least square means of the two groups. If the upper limit of the 95% confidence interval of the difference between the least square means of the main indicators is less than 0%, it indicates that the experimental group is superior to the control group.
2. Secondary efficacy measures: In this study, we assesse triglycerides, total cholesterol, high-density lipoprotein, non-high-density lipoprotein cholesterol, small-density low-density lipoprotein, low-density lipoprotein, Apolipoprotein. Protein B, tumor necrosis factor-alpha. The FAS set and the PPS set are used to compare the experimental and control groups. Percent change from baseline in LDL-C at months 1 and 6 will be assessed using statistical methods similar to those used for the primary outcome measure.
3. Security indicators: We use the chi-square test or Fisher's exact test to compare the incidence of adverse events and serious adverse events between the two groups, and tabulate all adverse events that occurred in this trial.

5.The total sample size of clinical trials and the reasons for their determination:

This clinical trial adopts a superiority test design. The experimental group and the control group are divided into groups according to 2:1. The main evaluation index is low-quality indicator. Describe as the percentage change from baseline in low-density lipoprotein cholesterol (LDL-C) in the experimental group or the control group at the 3rd month, respectively, the establishment of the hypothesis test is as follows:

Null hypothesis H0: T-C≥-∆; Alternative hypothesis H1: T-C<-∆; Among them, T and C are the least squares mean of the percentage change of low-density lipoprotein cholesterol relative to the baseline before treatment and 3 months of treatment in the experimental group and the control group, respectively, Δ is the superiority cutoff value, the superiority cutoff value of this trial Set to 0%.

When the superiority tests of the main evaluation indicators are all established, the superiority of this trial is established. Therefore no alpha correction is required.

Calculate the formula according to the sample size: According to the data of clinical literature, the LDL-C of subjects before and after drinking hydrogen water decrease by about 6%~18%, which is about 6~8% lower than that of placebo. Assuming that before treatment and after 3 months of treatment, the percentage difference between the experimental group and the control group in LDL-C from baseline is 6%, the standard deviation is 12%, the superiority margin is 0%, one-sided statistical test the significance level is 0.025, and the power is 80%. There are at least 95 cases in the experimental group and at least 48 cases in the control group. According to the 20% dropout rate, there are 120 cases in the test group and 60 cases in the control group, with a total of 180 cases.

6.Handling of missing data: Missing data are generally not filled, unless otherwise specified.

7.Minimum and maximum number of subjects and justification for each clinical trial facility: Due to the difference in the number of patients in each center, this trial will be conducted in a competitive manner among centers. For a given center, the final enrollment size should not be less than 10% of the total number of cases, and the maximum should not exceed 50% of the total number of cases.

8.Pass/Fail Criteria for Clinical Trial Results: Hypothesis testing of superiority is used in this clinical trial, and the main evaluation indicator is the percentage change from baseline in LDL cholesterol at 3 months of treatment. The superiority test is valid if the difference between the experimental group and the control group is less than 0% at the upper limit of the 95% confidence interval.

9.Statistical analysis software: This experiment will use SAS 9.4 or later for statistical analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 (inclusive), gender is not limited;
* Subjects with clinical diagnosis of hyperlipidemia;
* The subjects' fasting LDL-C and carotid artery color Doppler ultrasound meet one of the following requirements: 1. Bilateral carotid artery color Doppler shows no plaque formation, and 2.6 ≤ LDL-C < 4.92mmol/L; 2. Bilateral or unilateral neck Arterial plaque formation, and 2.6≤LDL-C<3.4mmol/L;
* 18.5 kg/m2≤BMI≤35 kg/m2, Body mass index (BMI) is calculated by dividing body weight (kg) by the square of height (m2);
* Subjects who are willing to participate in the trial and sign informed consent.

Exclusion Criteria:

* Secondary hyperlipidemia caused by systemic diseases (such as nephrotic syndrome, hypothyroidism, systemic lupus erythematosus, glycogen storage disease, liver disease or renal failure, etc.);
* Fasting triglycerides > 5.6 mmol/L;
* Diabetic patients;
* Those who plan to undergo bariatric surgery (gastric retraction, gastric bypass, gastric banding, etc.) during the study period;
* Have taken or plan to take lipid-lowering drugs within the last 8 weeks (eg, statins, cholesterol absorption inhibitors, probucol, bile acid sequestrants, fibrates, proprotein convertase subtilisin 9 (PCSK9) ) inhibitors, Xuezhikang and Chinese patent medicines with lipid-lowering effect, etc.) who intervene;
* Those who have taken or plan to take lipid-lowering drugs within the last 8 weeks (eg, statins, cholesterol absorption inhibitors, probucol, bile acid sequestrants, fibrates, proprotein convertase subtilisin 9 (PCSK9) inhibitors, Xuezhikang and Chinese patent medicines with lipid-lowering effect, etc.);
* Subjects who have used heparin, thyroxine treatment drugs, diuretics, phenothiazines, beta-blockers, adrenal corticosteroids and certain contraceptives in the past 8 weeks, which may affect blood lipid metabolism;
* Combined with malignant tumor or mental disorder;
* Accompanied by severe cardiovascular and cerebrovascular diseases, liver and kidney function damage (NYHA grade greater than or equal to 3, ALT or AST > 3 times the upper limit of normal, Cr > 1.5 times the upper limit of normal);
* Those who have participated in clinical trials of other drugs or medical devices within 3 months;
* Those who plan to become pregnant, are pregnant or are breastfeeding during the study period and those who cannot take contraceptive measures;
* Patients deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in LDL-C at 3 months of intervention. | At 3 months of intervention.
  LDL-C will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.

SECONDARY OUTCOMES:
Absolute change from baseline in LDL-C at 3 months of intervention. | At 3 months of intervention.
  LDL-C will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in LDL-C at 1 month of intervention. | at 1 month of intervention.
  LDL-C will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in LDL-C at 1 month of intervention. | at 1 month of intervention.
  LDL-C will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in LDL-C at 6 months of intervention. | at 6 months of intervention.
  LDL-C will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in LDL-C at 6 months of intervention. | at 6 months of intervention.
  LDL-C will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in triglycerides at 1 month of intervention. | At 1 month of intervention.
  Triglycerides will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in triglycerides at 1 month of intervention. | At 1 month of intervention.
  Triglycerides will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in triglycerides at 3 months of intervention. | At 3 months of intervention.
  Triglycerides will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in triglycerides at 3 months of intervention. | At 3 months of intervention.
  Triglycerides will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in triglycerides at 6 months of intervention. | At 6 months of intervention.
  Triglycerides will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in triglycerides at 6 months of intervention. | At 6 months of intervention.
  Triglycerides will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in total cholesterol at 1 month of intervention. | At 1 month of intervention.
  Total cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in total cholesterol at 1 month of intervention. | At 1 month of intervention.
  Total cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in total cholesterol at 3 months of intervention. | At 3 months of intervention.
  Total cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in total cholesterol at 3 months of intervention. | At 3 months of intervention.
  Total cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in total cholesterol at 6 months of intervention. | At 6 months of intervention.
  Total cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in total cholesterol at 6 months of intervention. | At 6 months of intervention.
  Total cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in HDL cholesterol at 1 month of intervention. | At 1 month of intervention.
  HDL cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in HDL cholesterol at 1 month of intervention. | At 1 month of intervention.
  HDL cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in HDL cholesterol at 3 months of intervention. | At 3 months of intervention.
  HDL cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in HDL cholesterol at 3 months of intervention. | At 3 months of intervention.
  HDL cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in HDL cholesterol at 6 months of intervention. | At 6 months of intervention.
  HDL cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in HDL cholesterol at 6 months of intervention. | At 6 months of intervention.
  HDL cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in non-HDL cholesterol at 1 month of intervention. | At 1 month of intervention.
  Non-HDL cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in non-HDL cholesterol at 1 month of intervention. | At 1 month of intervention.
  Non-HDL cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in non-HDL cholesterol at 3 months of intervention. | At 3 months of intervention.
  Non-HDL cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in non-HDL cholesterol at 3 months of intervention. | At 3 months of intervention.
  Non-HDL cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in non-HDL cholesterol at 6 months of intervention. | At 6 months of intervention.
  Non-HDL cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in non-HDL cholesterol at 6 months of intervention. | At 6 months of intervention.
  Non-HDL cholesterol will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in small and dense LDL at 1 month of intervention. | At 1 month of intervention.
  Small and dense LDL will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in small and dense LDL at 1 month of intervention. | At 1 month of intervention.
  Small and dense LDL will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in small and dense LDL at 3 months of intervention. | At 3 months of intervention.
  Small and dense LDL will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in small and dense LDL at 3 months of intervention. | At 3 months of intervention.
  Small and dense LDL will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in small and dense LDL at 6 months of intervention. | At 6 months of intervention.
  Small and dense LDL will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Absolute change from baseline in small and dense LDL at 6 months of intervention. | At 6 months of intervention.
  Small and dense LDL will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "mmol/L" as the unit.
Percent change from baseline in apolipoprotein B at 1 month of intervention. | At 1 month of intervention.
  Apolipoprotein B will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "g/L" as the unit.
Absolute change from baseline in apolipoprotein B at 1 month of intervention. | At 1 month of intervention.
  Apolipoprotein B will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "g/L" as the unit.
Percent change from baseline in apolipoprotein B at 3 months of intervention. | At 3 months of intervention.
  Apolipoprotein B will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "g/L" as the unit.
Absolute change from baseline in apolipoprotein B at 3 months of intervention. | At 3 months of intervention.
  Apolipoprotein B will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "g/L" as the unit.
Percent change from baseline in apolipoprotein B at 6 months of intervention. | At 6 months of intervention.
  Apolipoprotein B will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "g/L" as the unit.
Absolute change from baseline in apolipoprotein B at 6 months of intervention. | At 6 months of intervention.
  Apolipoprotein B will be uniformly implemented in the laboratories of each research central hospital.And uniformly use "g/L" as the unit.
Percent change from baseline in TNF-alpha at 1 month of intervention. | At 1 month of intervention.
  TNF-alpha will be uniformly implemented in the laboratories of each research central hospital. And uniformly use "pg/ml" as the unit.
Absolute change from baseline in TNF-alpha at 1 month of intervention. | At 1 month of intervention.
  TNF-alpha will be uniformly implemented in the laboratories of each research central hospital. And uniformly use "pg/ml" as the unit.
Percent change from baseline in TNF-alpha at 3 months of intervention. | At 3 months of intervention.
  TNF-alpha will be uniformly implemented in the laboratories of each research central hospital. And uniformly use "pg/ml" as the unit.
Absolute change from baseline in TNF-alpha at 3 months of intervention. | At 3 months of intervention.
  TNF-alpha will be uniformly implemented in the laboratories of each research central hospital. And uniformly use "pg/ml" as the unit.
Percent change from baseline in TNF-alpha at 6 months of intervention. | At 6 months of intervention.
  TNF-alpha will be uniformly implemented in the laboratories of each research central hospital. And uniformly use "pg/ml" as the unit.
Absolute change from baseline in TNF-alpha at 6 months of intervention. | At 6 months of intervention.
  TNF-alpha will be uniformly implemented in the laboratories of each research central hospital. And uniformly use "pg/ml" as the unit.
Adverse Event (AE) Frequency | At 6 months of intervention.
  Record the Adverse Event (AE) Frequency, compare the AE between two groups using chi square test or Fisher's exact probability method, and list all AE that occurred in this trial.
Severe Adverse Event (SAE) Frequency | At 6 months of intervention.
  Record the Severe Adverse Event (SAE) Frequency, compare the SAE between two groups using chi square test or Fisher's exact probability method, and list all SAE that occurred in this trial.
Device deficiency rate | At 6 months of intervention.
  Record the device deficiency rate, measure the stability evaluation of device.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Sun, MD,PhD, Study Chair — Zhujiang Hospital; Hong Chen, MD,PhD, Principal Investigator — Zhujiang Hospital; Li Cong, MD,PhD, Principal Investigator — Fifth Affiliated Hospital, Sun Yat-Sen University; Lihong Wang, MD,PhD, Principal Investigator — First Affiliated Hospital of Jinan University; Xiuwei Zhang, MD,PhD, Principal Investigator — Dongguan People's Hospital; Yi Shu, MD,PhD, Principal Investigator — Foshan Nanhai District People's Hospital
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No